CLINICAL TRIAL: NCT01544530
Title: Feasibility of Mild-to-moderate Therapeutic Hypothermia as an In-vivo Organ Preservation Strategy in Brain-dead Donors
Brief Title: Cooling to Optimize Organ Life in Donor Study
Acronym: COOLDonor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding and other logistic reasons
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Raghavan Murugan, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORID - 335
Record Dates: First submitted 2011-11-21; First posted 2012-03-06 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Organ Transplantation From Brain-dead Donors
Keywords: Brain-death; organ donation
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia (32-33 degree C) (Experimental): Following randomization, hypothermia will be induced by a combination of cold isotonic fluid and sustained until organ procurement by a central venous catheter
  Interventions: Other: Cold isotonic fluid and central venous hypothermia catheter
- Normothermia (36.5 - 37.5 degree C) (No Intervention): Normothermia will be maintained until organ procurement as per current standard of care

INTERVENTIONS:
Other: Cold isotonic fluid and central venous hypothermia catheter — 20-30ml/kg of isotonic crystalloid resuscitation fluid will be used for induction. Hypothermia (32-33 degrees C) will be sustained until organ procurement using an FDA approved central venous catheter connected to an external temperature regulating system
  Arms: Hypothermia (32-33 degree C)

SUMMARY:
The purpose of this study is to assess the feasibility and safety of mild-to-moderate hypothermia as an in-vivo organ preservation strategy compared to normothermia in 60 brain-dead organ donors.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years;pronounced dead as per hospital brain-death criteria
* Accepted by organ procurement organization for organ donation
* Subjects within 3 hours of brain death pronouncement

Exclusion Criteria:

* Consent cannot be obtained from authorized representative;mean arterial pressure < 60 mmHg and/ or more than 2 vasopressor and/or inotrope use
* Presence of 2nd or 3rd degree heart block
* Ongoing extracranial hemorrhage
* International normalized ratio > 3.0
* Donors with human-immunodeficiency virus infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety | From enrollment to organ procurement (average of 24 hours)
  Brain-dead organ donors will be followed from study enrollment up to organ procurement for an average of 24 hours

SECONDARY OUTCOMES:
Six-month hospital free survival in recipients | 6 months
  Data on recipient survival and allograft function will be collected up to 6 months following transplantation
Interleukin-6 | Baseline, 6 hours, and at organ procurement (15-24 hrs)
Actual no. of organs transplanted | At the time of organ procurement
Malondialdehyde | Baseline, 6 hours, and at organ procurement (15-24 hrs)
Death receptor-5 | Baseline, 6 hours, and at organ procurement (15-24 hrs)
lactate | Baseline, 6 hours, and at organ procurement (15-24 hrs)
Urinary isoprostanes | Baseline, 6 hours, and at organ procurement (15-24 hrs)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States